CLINICAL TRIAL: NCT05496556
Title: Influence of Food Preferences on the Occurrence of Undernutrition in Treated Patients for Bronchopulmonary Carcinoma Non-small Cell Stage IV
Acronym: ONCOGOU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A01952-39
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Bronchopulmonary Carcinoma at Stage IV and Benefiting From First-line Treatment According to Current French Recommendations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients included in the study (Other): Patient with stage IV non-small cell bronchopulmonary carcinoma receiving first-line treatment and received LFQP questionnaire
  Interventions: Other: Test Leeds Food Preference Questionnaire (LFQP-France)

INTERVENTIONS:
Other: Test Leeds Food Preference Questionnaire (LFQP-France) — The version of this questionnaire has been adapted to French eating habits. and based on the presentation of food photos, each representing one of the four categories below : salty-high in fat / salty-low fat / sugary-high fat / sweet-low fat The answers given to the LFQP predict a more or less caloric food intake. This tool makes it possible to objectify changes in eating behavior according to the nutritional status and protein status of patients.
  The implied wanting score for salty-high-fat, salty-low-fat, sweet-high-fat, and sweet-low-fat foods is calculated based on the frequency and speed of choice for one food type out of 150 combinations.
  For each of the food modalities, the software will return a score with its standard deviation. The modality preferred by the patient is the one with the highest score

SUMMARY:
The study will be offered to patients with non-small cell lung carcinoma diagnosed at stage IV and receiving first-line treatment.

The patient will benefit from a complete assessment at inclusion (clinical exam, imagery, biological exam, dietary consultation, test LFQP.

At the end of this 1st evaluation, patients in whom the diagnosis of undernutrition is made will benefit from dietary management with personalized advice that will take into account the symptoms of cancer, the possible side effects of treatments as well as the social environment.

Every two cures, i.e. every 4 to 6 weeks, these examens will be performed until the occurrence of an event (progression of the disease according to the RECIST criteria, death or change of therapeutic line). At the end of these assessments, patients will benefit from dietary management with a readjustment of personalized advice that will take into account the difficulties highlighted during the assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV non-small cell lung carcinoma with indication for first-line systemic treatment (chemotherapy, immunotherapy or specific treatment, in particular tyrosine kinase inhibitors) according to current French recommendations.
* Age over 18 and under 70
* Patient speaking and reading French fluently
* Affiliation to a social security scheme
* Patient able and willing to follow all study procedures in accordance with the protocol
* Patient having understood, signed and dated the consent form

Exclusion Criteria:

* Patient requiring hospitalization for more than 48 hours for the administration of the first course of treatment
* Patient benefiting from antibiotic therapy for the treatment of an acute infection
* Psychiatric, cognitive or neurological disorders making it impossible to assess food preferences and/or any impossibility to undergo medical monitoring for the trial for geographical, social or psychological reasons.
* Daily alcohol consumption
* Chest radiotherapy treatment
* Pregnant woman, likely to be, or breastfeeding
* Persons deprived of liberty or under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of implicit wanting by the LFQP-France questionnaire | During patient follow-up (12 months max)
  The food category with the highest implicit wanting score will be retained as characterizing the patient's food preferences. The 4 categories concerned are as follows:
  * salty high in fat
  * salty-low fat
  * sweet-high fat
  * sweet-low fat

SECONDARY OUTCOMES:
The occurrence of undernutrition within 6 months after inclusion, in patients not undernourished at inclusion | During 6 months
  The food category with the highest implicit wanting score will be retained as characterizing the patient's food preferences. The 4 categories concerned are as follows:
  * salty high in fat
  * salty-low fat
  * sweet-high fat
  * sweet-low fat
The impact of food preferences (liking and explicit wanting) assessed by the LFQP-France questionnaire on the prevalence and incidence of undernutrition in the 6 months after inclusion. | During 6 months
  The food category with the highest implicit wanting score will be retained as characterizing the patient's food preferences. The 4 categories concerned are as follows:
  * salty high in fat
  * salty-low fat
  * sweet-high fat
  * sweet-low fat
The impact of food preferences (liking, explicit lwanting and implicit wanting) assessed by the LFQP-France questionnaire on the severity of undernutrition | through study completion, an average of 1 year
  The severity of malnutrition will be determined by serum albumin.
the impact of food preferences (liking, explicit wanting and implicit wanting) assessed by the LFQP-France questionnaire on quality of life | through study completion, an average of 1 year
  With the EORTC QLQ-C30 and QLQ-CL13 tests at inclusion, then at each follow-up visit and until exit from the study (premature exit or end of study
The impact of the type of 1st line treatment on food preferences (chemotherapy based on platinum salt versus immunotherapy versus targeted therapy) | through study completion, an average of 1 year
  1st line treatments considered categorized into 3 classes: platinum-based chemotherapy versus immunotherapy versus targeted therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges-François Leclerc, Dijon, Côte d'Or, France